CLINICAL TRIAL: NCT06435364
Title: Investigation of the Effect of Instrument Supported Cervical Manual Therapy Methods and Vagus Nerve Stimulation in Patients With Nonspecific Neck Pain
Brief Title: Cervical Manual Therapy and Vagus Nerve Stimulation in Patients With Nonspecific Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-2983
Record Dates: First submitted 2024-05-24; First posted 2024-05-30 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Pain Syndrome
MeSH Terms: conditions — Somatoform Disorders | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vagus nerve (Experimental): This non-invasive system is activated by the cutaneous distribution of vagus nerve afferents via the external ear.
  Interventions: Other: Vagus nerve stimilation
- Manual therapy (Active Comparator): Manual therapy is effective in the treatment of musculoskeletal pain.
  Interventions: Other: Manual therapy

INTERVENTIONS:
Other: Vagus nerve stimilation — This non-invasive system is activated by the cutaneous distribution of vagus nerve afferents through the external ear. Somatosensory innervation is provided by the auricular branch.
  Arms: Vagus nerve
Other: Manual therapy — Manual therapy is mostly defined by the tissue targeted by the practitioner; it can be joint biased, muscle and connective tissue biased and/or neurovascular system biased techniques.
  Arms: Manual therapy

SUMMARY:
People with chronic neck pain are becoming more and more common in society every day.

DETAILED DESCRIPTION:
In chronic neck pain investigations, it is generally reported that all people experience neck pain once in my life and more than half of the developed societies experience this problem. It has been stated that 48% of these continue as chronic neck pain, which significantly affects the quality of life due to the postponement of treatment due to its cost.

ELIGIBILITY:
Inclusion criteria for volunteers and/or study participants;

* Presence of neck pain for at least three months
* Non-specific neck pain
* To have signed the voluntary consent form

Exclusion criteria for volunteers and/or participants;

* Having undergone surgery for the cervical region
* Rehabilitation of the neck area at least three months prior to treatment
* Traumatic medulla spinalis injury
* Neurological deficit
* Rheumatological disease
* Structural spinal disorders

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-05-17 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-08-21 (Actual)

PRIMARY OUTCOMES:
Heart rate variability | 4 weeks
  Heart rate variability (HRV) is an indicator of the effects of these two components on the heart, reflecting the variations in the time intervals between heartbeats. High HRV generally indicates good autonomic balance and a healthy cardiovascular system, while low HRV can be a sign of stress, fatigue, or underlying health issues. When sympathetic nervous system activity increases, heart rate accelerates and HRV decreases; conversely, when parasympathetic nervous system activity increases, heart rate slows and HRV increases. Therefore, HRV is an important biomarker for assessing overall health status and developing stress management strategies.
Neck disability index: | 4 weeks
  The neck disability index is the most commonly used functional outcome tool for disabilities in the cervical region. This outcome assessment tool was created by modifying the Oswestry Disability Index and is highly reliable (Chad E. Cook, Amy E. Cook 2011).
  Scoring is given for each question as A: 0 points, B: 1 point, C: 2 points, D: 3 points, E: 4 points, F: 5 points. The total score gives the test score. According to the test result 0-4=No disability 5-14= Mild disability 15-24= Moderate disability 25-34 = Severe disability
Joint Range of Motion | 4 weeks
  Range of motion is the ability of a joint to go through the full range of motion. The range of motion of a joint can be passive or active. Passive ROM - The maximum range of motion through which the joint can move with the aid of external force. Active ROM - the range of motion achieved by contracting and relaxing opposing muscles
The visual analogue scale (VAS) | 4 weeks
  The visual analogue scale (VAS) is a validated, subjective measure of acute and chronic pain. Scores are recorded by placing a handwritten mark on a 10 cm line representing the continuum between "no pain" and "worst pain"

CONTACTS AND LOCATIONS:
Locations (1):
- Bahçehir University, Istanbul, Turkey (Türkiye)